CLINICAL TRIAL: NCT06656234
Title: The Effectiveness and Safety of Glofitamab in Real-World Clinical Practice Among Chinese Adult Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma: A Prospective, Observational, Multicenter Study
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Prof., Ruijin Hospital
Other Study IDs: GloReal
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — glofitamab; obinutuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with relapsed or refractory (R/R) DLBCL who have started receiving glofitamab at physician's discretion in accordance with local clinical practice and/or labeling will be observed for safety and efficacy until death, withdrawal of consent, loss to follow-up or end of study whichever occurs first (up to approximately 4 years).
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Glofitamab — Glofitamab will be administered at the discretion of the physician per local clinical practice and local labeling.
Drug: Obinutuzumab — Obinutuzumab pre-treatment is given intravenously at a dose of 1g on Cycle 1 Day 1.

SUMMARY:
The purpose of this study is to evaluate the the efficacy and safety in the real-world settings of glofitamab among Chinese R/R DLBCL participants.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed as R/R DLBCL
* Participants who will be treated with glofitamab (known as being recommended and having the intention to be treated with glofitamab at the time of signing informed consent) or have initiated glofitamab treatment within 6 months prior to enrollment and after the indication approval will be observed in this study.

Exclusion Criteria:

* Any other reason that, in the investigator's opinion, makes the participant unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who will be treated with glofitamab (known as being recommended and having the intention to be treated with glofitamab at the time of signing informed consent) or have initiated glofitamab treatment within 6 months prior to enrollment and after the indication approval will be observed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | Baseline up to end of study (EOS) (approximately 48 months)

SECONDARY OUTCOMES:
Complete Response Rate (CRR) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | Baseline up to EOS (approximately 48 months)
Overall Response Rate (ORR) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | Baseline up to EOS (approximately 48 months)
Duration of Response (DoR) | From the date of the first occurrence of a documented CR or partial response (PR) to the date of progression, relapse, or death from any cause, whichever occurs first (up to approximately 48 months)
Duration of Complete Response (DoCR) | From the date of the first occurrence of a documented CR to the date of progression, relapse, or death from any cause, whichever occurs first (up to approximately 48 months)
Time to Next Treatment (TTNT) | From the start of glofitamab treatment to the initiation of next-line treatment (up to approximately 48 months)
Overall Survival (OS) | From the start of glofitamab treatment until the date of death from any cause (up to approximately 48 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No